CLINICAL TRIAL: NCT06467266
Title: Mechanistic Insights From Multisite Pacing in Patients With Heart Failure With Preserved Ejection Fraction
Brief Title: Mechanistic Insights From Temporary Pacing in HFpEF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 332571
Record Dates: First submitted 2024-06-05; First posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Heart Failure Preserved Ejection Fraction; Pacing
MeSH Terms: conditions — Heart Failure, Diastolic

STUDY DESIGN:
Intervention Model Description: This is an observational cohort mechanistic study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Patients will undergo cardiac imaging with a cardiac MRI and echocardiogram prior to the haemodynamic study. The haemdynamic study will be performed in the catheter lab. During that study patients will undergo a temporary pacing procedure with pacing of multiple sites of the heart and multiple haemodynamic recordings. This will be conducted under local anaesthetic and sedation. Total procedure time will be approximately 2 hours.
  Interventions: Diagnostic Test: Acute Haemodynamic Study

INTERVENTIONS:
Diagnostic Test: Acute Haemodynamic Study — Multisite temporary pacing

SUMMARY:
Heart failure with preserved ejection fraction (HFpEF) is characterised by impaired diastolic function. A recent clinical trial has demonstrated multiple beneficial outcomes in HFpEF patients receiving personalised accelerated pacing from indwelling permanent pacemakers, including symptomatic improvement, objective reductions in NT-proBNP level and AF-burden.

The investigators aim to determine the underlying mechanisms behind these documented effects, to investigate the acute intracardiac haemodynamic response to temporary multisite pacing in HFpEF participants and to gain further mechanistic insight with additional haemodynamic, electrical and echocardiographic data collection during temporary pacing in this cohort. This will all provide valuable information towards new potential targets of therapy.

DETAILED DESCRIPTION:
In this research study, the investigators will perform a one-off temporary pacing procedure in the catheter lab at St Thomas' Hospital in patients with heart failure with preserved ejection fraction (HFpEF). During the short procedure, the investigators will pace the heart at different heart rates and from different parts of the heart. The investigators will measure the change in pressure inside the heart in response to each pacing site/mode and rate. Altogether, the investigators aim to find out how different pacing modes and heart rates impact how well the heart fills and pumps in HFpEF.

The study will provide valuable information about the underlying mechanisms of pacing in HFpEF, which could significantly influence the future direction of HFpEF management. Specifically, it will help the investigators to understand what types of pacemaker and pacing site or pacing mode may be chosen in HFpEF patients requiring pacing, which accounts for around 20% of all HFpEF patients.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* Formal diagnosis of HFpEF as per ESC guidelines
* NYHA grade II-IV heart failure symptoms
* LVEF ≥50%
* Female participants of child-bearing potential must be willing to ensure that they or their partner use effective contraception during the study and for 3 months thereafter
* Able (in the Investigators opinion) and willing to comply with all study requirements.
* Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the study.

Exclusion Criteria:

* History of persistent or permanent AF
* Permanent pacing device in situ
* Female participants who are pregnant, lactating or planning pregnancy during the course of the study.
* Scheduled elective surgery or other procedures requiring general anaesthesia during the study.
* Participant who is terminally ill
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
* Significant peripheral vascular disease precluding an EP study
* A contraindication to anticoagulation
* A prosthetic aortic, mitral or tricuspid valve
* Significant Aortic valve disease
* Known LV thrombus
* Insufficient capacity to consent to the study
* Participation in other studies with active treatment / investigational arm to avoid bias

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with changes in left ventricular end diastolic pressure upon accelerated right atrial pacing and conduction system pacing | 30 months
  Measurement of the absolute left ventricular end diastolic pressure (in mmHg) and volume (in milliliter) at real-time during each pacing mode, heart rate and AV delay with a pressure volume loop catheter

SECONDARY OUTCOMES:
Number of participants with leftward, downward shift in the LV P-V loop during accelerated RA pacing and CSP, not reproduced by RV pacing | 30 months
  Qualitative assessment of the leftward, downward shift in the left ventricular P-V loop during accelerated right atrial pacing and conduction system pacing, not reproduced by right ventricular pacing
Number of participants with changes in Echo measures of diastology upon right atrial pacing and conduction system pacing | 30 months
  Measurement of the absolute left ventricular tissue velocity (measured in centimeter/second) with the use of a pulse wave tissue doppler imaging (TDI) signal in the apical four chamber view

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Infeld M, Wahlberg K, Cicero J, Plante TB, Meagher S, Novelli A, Habel N, Krishnan AM, Silverman DN, LeWinter MM, Lustgarten DL, Meyer M. Effect of Personalized Accelerated Pacing on Quality of Life, Physical Activity, and Atrial Fibrillation in Patients With Preclinical and Overt Heart Failure With Preserved Ejection Fraction: The myPACE Randomized Clinical Trial. JAMA Cardiol. 2023 Mar 1;8(3):213-221. doi: 10.1001/jamacardio.2022.5320. PMID 36723919
- [Background] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2021 Sep 21;42(36):3599-3726. doi: 10.1093/eurheartj/ehab368. No abstract available. PMID 34447992
- [Background] Reddy YNV, Koepp KE, Carter R, Win S, Jain CC, Olson TP, Johnson BD, Rea R, Redfield MM, Borlaug BA. Rate-Adaptive Atrial Pacing for Heart Failure With Preserved Ejection Fraction: The RAPID-HF Randomized Clinical Trial. JAMA. 2023 Mar 14;329(10):801-809. doi: 10.1001/jama.2023.0675. PMID 36871285
- [Background] Elliott MK, Strocchi M, Sieniewicz BJ, Sidhu B, Mehta V, Wijesuriya N, Behar JM, Thorpe A, Martic D, Wong T, Niederer S, Rinaldi CA. Biventricular endocardial pacing and left bundle branch area pacing for cardiac resynchronization: Mechanistic insights from electrocardiographic imaging, acute hemodynamic response, and magnetic resonance imaging. Heart Rhythm. 2023 Feb;20(2):207-216. doi: 10.1016/j.hrthm.2022.10.019. Epub 2022 Oct 28. PMID 36575808
- [Background] Dunlay SM, Roger VL, Redfield MM. Epidemiology of heart failure with preserved ejection fraction. Nat Rev Cardiol. 2017 Oct;14(10):591-602. doi: 10.1038/nrcardio.2017.65. Epub 2017 May 11. PMID 28492288